CLINICAL TRIAL: NCT02850952
Title: Rehab MATRIX: Impact of a Nursing-Led Acuity Algorithm on Patient Safety and Healthcare Quality
Acronym: Rehab MATRIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Texas Medical Center (Unknown); Memorial Hermann Health System (Other)
Responsible Party: Principal Investigator, Nneka Lotea Ifejika, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HSC-MS-16-0358
Record Dates: First submitted 2016-07-21; First posted 2016-08-01 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Nurse's Role; Nurse-Patient Relations; Satisfaction; Patient Fall
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rehab MATRIX (Experimental): Rehab MATRIX is a patient assignment tool that objectively categorizes patients undergoing inpatient rehabilitation based on nurse identified acuity variables.
  Interventions: Other: Rehab MATRIX

INTERVENTIONS:
Other: Rehab MATRIX — Rehab MATRIX is a patient assignment tool that objectively categorizes patients undergoing inpatient rehabilitation based on nurse identified acuity variables.

SUMMARY:
To determine whether implementation of Rehab MATRIX will improve patient safety, patient satisfaction and nursing indices.

DETAILED DESCRIPTION:
The provision of efficient and conscientious nursing care is at the forefront of health care quality. Unfortunately, a lack of objectivity in the assignment of patients to nurses can lead to inequalities of care. Such inequalities translate to poor patient outcomes and diminished patient satisfaction. Furthermore, staff attrition related to nursing fatigue increases the cost of care due to a reliance on supplemental nurses. Rehab MATRIX is a patient assignment tool that objectively categorizes patients undergoing inpatient rehabilitation based on nurse identified acuity variables.

ELIGIBILITY:
Inclusion Criteria:

* Rehabilitation Nursing Staff within Six Study Centers
* Patient hospitalized within the Rehabilitation Unit during the study period

Exclusion Criteria:

* Other Nursing Staff
* Patients hospitalized on non-rehabilitation units

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in the number of falls per 1000 patient days (falls per 100 patient days is a standardized proportion) | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months

SECONDARY OUTCOMES:
Change in Patient Satisfaction as assessed by the Press Ganey Survey | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
Change in Nursing Fatigue as assessed by number of unexcused nurse absences | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months
Change in Nursing Satisfaction as assessed by a survey | Two weeks prior to initiation, 6 months
  Two weeks prior to Rehab MATRIX initiation, a six question pre-implementation survey will be distributed via Survey Monkey to the nursing staff, evaluating nurse perceptions of the traditional nursing assignment. Questions 1 to 4 will be measured on a Likert Scale of 1 to 5; 1 - strongly disagree, 2 - disagree, 3 - neutral, 4 - agree, 5 - strongly agree.
  At the end of the six month study period, a post-implementation Rehab MATRIX survey will be distributed at each center via Survey Monkey, examining the impact of Rehab MATRIX on workload equity, fairness, the role of seniority and overall satisfaction with the nurse assignment process.

CONTACTS AND LOCATIONS:
Overall Officials: Nneka L Ifejika, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Result] Ifejika NL, Okpala MN, Moser HA, Watkins JN, Noser EA. Rehab MATRIX: Content Validity of a Nursing-Led Patient Assignment Algorithm. J Neurosci Nurs. 2019 Feb;51(1):33-36. doi: 10.1097/JNN.0000000000000418. PMID 30614934